CLINICAL TRIAL: NCT00631449
Title: Raltegravir Intensification in Antiretroviral-treated Patients Exhibiting a Suboptimal CD4+ T Cell Response
Brief Title: Raltegravir Intensification in HIV-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H52899-31393-03
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: HIV Infections
Keywords: HIV; Treatment intensification; Low level viremia; Suboptimal CD4+ T cell response; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir (Active Comparator): For subjects assigned to the raltegravir group, subjects will receive raltegravir 400 mg to be taken by mouth twice daily for 24 weeks, in addition to continuing to take their current anti-HIV medicines.
  Interventions: Drug: Raltegravir
- Placebo (Placebo Comparator): For subjects assigned to the placebo group, subjects will receive a matching placebo pill 400 mg to be taken by mouth twice daily for 24 weeks, in addition to continuing to take their current anti-HIV medicines.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raltegravir — For subjects assigned to the raltegravir group, subjects will receive raltegravir 400 mg to be taken by mouth twice daily, in addition to continuing to take their current anti-HIV medicines.
  Arms: Raltegravir
Drug: Placebo — For subjects assigned to the placebo group, subjects will receive a matching placebo pill 400 mg to be taken by mouth twice daily for 24 weeks, in addition to continuing to take their current anti-HIV medicines.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treatment with Raltegravir further decreases HIV viral replication in HAART-suppressed, HIV-infected patients, potentially improving immune response to antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Stable antiretroviral therapy for at least 12 months
* Screening CD4+ T cell count < 350 cells/mm3
* All available CD4+ T cell counts in the last year and at screening < 350 cells/mm3
* Screening plasma HIV RNA levels below level of detection (< 50 copies RNA/mL using Roche Amplicor or < 75 copies/mL using Bayer bDNA or < 40 copies/mL using Abbott RT-PCR), and all available determinations in past 12 months also below level of detection (isolated single values > 75 but < 1000 copies/mL will be allowed if they were preceded and followed by undetectable viral load determinations).
* >90% adherence to therapy within the preceding 30 days, as determined by self-report
* Both male and female adult (at least 18 years old) subjects are eligible. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.

Exclusion Criteria:

* Patients who are intending to modify antiretroviral therapy in the next 24 weeks for any reason
* Serious illness requiring hospitalization or parental antibiotics within preceding 3 months
* **Any vaccination 2 weeks prior to baseline (day 0) visit and throughout the study period
* Concurrent treatment with immunomodulatory drugs, or exposure to any immunomodulatory drug in past 16 weeks
* Concurrent treatment with phenobarbital, phenytoin, or rifampin.
* Screening absolute neutrophil count <1,000 cells/mm3, platelet count <70,000 cells/mm3, hemoglobin < 8 mg/dL, estimated creatinine clearance <40 mL/minute
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco General Hospital, Clinical Research Center, San Francisco, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California

REFERENCES:
- [Result] Hatano H, Hayes TL, Dahl V, Sinclair E, Lee TH, Hoh R, Lampiris H, Hunt PW, Palmer S, McCune JM, Martin JN, Busch MP, Shacklett BL, Deeks SG. A randomized, controlled trial of raltegravir intensification in antiretroviral-treated, HIV-infected patients with a suboptimal CD4+ T cell response. J Infect Dis. 2011 Apr 1;203(7):960-8. doi: 10.1093/infdis/jiq138. PMID 21402547

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raltegravir | Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (10.3) | 51.2 (8.0) | 51.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Group (Study Drug vs. Placebo) With Undetectable Plasma HIV-1 RNA, as Measured by an Ultra-sensitive Assay With a Limit of Detection of 1 Copy/mL at Week 12.
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Raltegravir | Placebo
Number analyzed (Participants) | 15 | 15
participants | 11 | 8

2. Secondary Outcome: Change in Percentage of Activated CD8+ T Cells (CD8+ T Cells That Co-express CD38 and HLA-DR) From Baseline to Week 24
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: Percentage of Activated CD8+ T cells
Arm/Group | Raltegravir | Placebo
Number analyzed (Participants) | 15 | 15
Percentage of Activated CD8+ T cells | -1.1 (NA) — PI has left the institution, the only access to the data is the publication and no data for measure of dispersion are available. | -0.9 (NA) — PI has left the institution, the only access to the data is the publication and no data for measure of dispersion are available.

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Raltegravir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No